CLINICAL TRIAL: NCT01709253
Title: Phase 2 Hypofractionation Study Using Proton Beam Therapy for Prostate Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Kwan Ho Cho, M.D., National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS 07-253
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Prostate Adenocarcinoma
Keywords: hpofractionation study using proton beam therapy
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): 27pt/60CGE/20fx/5wks to PGTV(mon, tue, thu, fri; 4/wk)
  Interventions: Radiation: proton beam therapy
- Arm 2 (Experimental): 27pt/54CGE/15fx/5wks to PGTV (mon, wed, fri; 3/wk)
  Interventions: Radiation: proton beam therapy
- Arm 3 (Experimental): 27pt / 47CGE/10fx/5wk to PGTV(tue, thu;2/wk)
  Interventions: Radiation: proton beam therapy
- Arm 4 (Experimental): 27pt/ 35CGE/ 5fx/2.5wk to PGTV(the, thu; 2/wk)
  Interventions: Radiation: proton beam therapy

INTERVENTIONS:
Radiation: proton beam therapy — hypofractionation study using proton beam therapy for prostate adenocarcinoma

SUMMARY:
Phase 2 hypofractionation study usion proton beam therapy for prostate adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

Biopsy proven prostate adenocarcinoma Stage: T1-T2cN0M0 ECOG performance status: 0-2 Signed study specific informed consent prior to study entry

Exclusion Criteria:

Postoperative residual or recurrent tumor Evidence of distant metastases Previous irradiation for the tumor in the same location Adjuvant anti-androgenic hormonal therapy High risk group (NCCN guide line)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
clinical outcomes | up to 5years from a initial follow-up
  To evaluate biochemical failure-free survival (BCFFS)

SECONDARY OUTCOMES:
acute toxicity | up to 5years from a initial follow-up
  to evaluate acute toxicities by CTCAE version 3.0
late toxicity | up to 5years from a initial follow-up
  to evaluated late toxicities by CTCAE version 3.0
overall survival | up to 5years from a initial follow-up
  to evaluated overall survival

CONTACTS AND LOCATIONS:
Overall Officials: kwan ho cho, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National cancer center, korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Ha B, Cho KH, Lee KH, Joung JY, Kim YJ, Lee SU, Kim H, Suh YG, Moon SH, Lim YK, Jeong JH, Kim H, Park WS, Kim SH. Long-term results of a phase II study of hypofractionated proton therapy for prostate cancer: moderate versus extreme hypofractionation. Radiat Oncol. 2019 Jan 10;14(1):4. doi: 10.1186/s13014-019-1210-7. PMID 30630500